CLINICAL TRIAL: NCT05489692
Title: Hepatic Arterial Infusion Chemotherapy Plus Targeted Therapy and/or PD-1 Inhibitors as Conversion Treatment for Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: HAIC Plus Targeted Therapy and/or PD-1 Inhibitors for Unresectable Intrahepatic Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Other Study IDs: B2022-222-01
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Hepatic Arterial Infusion Chemotherapy; Targeted Therapy; PD-1 Inhibitors
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Folfox protocol; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FOLFOX-HAIC plus targeted therapy and/or PD-1 inhibitors: FOLFOX-HAIC as the following dosage: 130 mg/m2 oxaliplatin infusion for 2 hours; 400 mg/m2 of leucovorin infusion for 2 hours; and 400 mg/ m2 of 5-FU bolus and 1200 of mg/m2 continuous infusion of 5-FU for 23 hours.
  Patients received targeted therapy, three different targeted therapy were applied including: 1. lenvatinib 2. sorafenib; 3. apatinib. A portion of patients received PD-1 inhibitor administered intravenously every three weeks.
  Interventions: Procedure: hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, fluorouracil, and leucovorin (FOLFOX)

INTERVENTIONS:
Procedure: hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, fluorouracil, and leucovorin (FOLFOX) — FOLFOX-HAIC as the following dosage: 130 mg/m2 oxaliplatin infusion for 2 hours; 400 mg/m2 of leucovorin infusion for 2 hours; and 400 mg/ m2 of 5-FU bolus and 1200 of mg/m2 continuous infusion of 5-FU for 23 hours.
  Patients received targeted therapy, three different targeted therapy were applied including: 1. lenvatinib 2. sorafenib; 3. apatinib. A portion of patients received PD-1 inhibitor administered intravenously every three weeks.
  Other Names: targeted therapy; PD-1 inhibitors

SUMMARY:
Intrahepatic cholangiocarcinoma (ICC) is associated with poor prognosis. This study aims to explore the efficacy and safety FOLFOX-HAIC in combination with targeted therapy and/or PD-1 inhibitors for patients with initially unresectable ICC, as well as its role in conversion therapy. Data were retrospectively reviewed for patients with locally advanced unresectable ICC treated with FOLFOX-HAIC combined with targeted therapy and/or PD-1 inhibitors. The treatment efficacy and safety were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were initially diagnosed without any previous oncological treatment.
2. The tumor was assessed as unresectable by two hepatobiliary surgeons (BL and YY, with more than 15 years of experience). Any of the following conditions: (1) Residual liver volume less than 30-40%; (2) Not possible for R0 radical resection; (3) Tumor invades the portal vein, hepatic artery and bile duct, and the normal residual liver cannot be guaranteed blood supply and bile drainage; the tumor involves the hepatic veins and cannot preserve at least one vein.
3. At least one assessable intrahepatic lesion.
4. classified as Child-Pugh Grade A.
5. ECOG PS score 0-1.
6. baseline blood tests meet the following criteria: leukocytes ≥3.0×10^9/L; neutrophils ≥1.5×10^9/L; platelets ≥75×10^9/L; hemoglobin ≥ 80g/L; serum ALT or AST ≤ 3 times of upper limit of normal (ULN); serum creatinine ≤1.5 x ULN; INR ≤ 1.5, or prothrombin time ≤ ULN + 4 seconds; albumin ≥ 30 g/L; total bilirubin ≤ 3 x ULN.

Exclusion Criteria:

1. severe underlying cardiac, pulmonary, or renal diseases.
2. a second primary malignancy.
3. prior history of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We reviewed data of patients diagnosed as ICC according to pathology or typical imaging presentation with elevated CA-199 between September 2017 and October 2021 at Sun Yat-Sen University Cancer Center. Patients with ICC confined to the liver and/or regional lymph nodes and treated by FOLFOX-HAIC combined with targeted therapy and anti-PD-1 therapy were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Tumor Response | 12 months
  The tumor responses were evaluated by measuring the longest diameter of target lesions according to response evaluation criteria in solid tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall survival (OS) was measured from the initiation of transarterial therapy to the date of death or the last follow-up.
Progression-free survival | 24 months
  Progression-free survival (PFS) was measured from the initiation of transarterial therapy to the time of progression or recurrence or last follow-up.
Conversion rate | 24 months
  Rate of patients underwent hepatic surgery after careful evaluation when an estimated residual liver volume >30-40% could be remained after R0 surgery by 2 experienced surgeons.

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No